CLINICAL TRIAL: NCT06070506
Title: Deep Learning-Based Prediction Model of Heart Failure With Improved Ejection Fraction
Brief Title: Heart Failure With Improved Ejection Fraction and Deep Learning
Status: Completed | Type: Observational
Sponsor: Yihui Kong (Other)
Responsible Party: Sponsor-Investigator, Yihui Kong, Professor, First Affiliated Hospital of Harbin Medical University
Organization: First Affiliated Hospital of Harbin Medical University (Other)
Other Study IDs: 2020020668
Record Dates: First submitted 2023-08-30; First posted 2023-10-06 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Heart Failure; Diagnosis
Keywords: Heart failure; Left ventricular ejection fraction; Heart failure with improved ejection fraction; Deep learning
MeSH Terms: conditions — Heart Failure; Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HFrEF group: Heart failure patients with LVEF persistently ≤40%.
- HFimpEF group: Heart failure patients with previous LVEF ≤40% and a follow-up LVEF of more than 40%.

SUMMARY:
The aim of this study was to design a deep learning-based trained model to assist in HFimpEF diagnosis.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years.
2. The diagnostic criteria of HF follows the 2018 Chinese Guidelines for the Diagnosis and Treatment of Heart Failure, having symptoms of dyspnea, fatigue or decreased activity tolerance, having signs of fluid retention (such as pulmonary congestion and peripheral edema), having echocardiogram abnormalities in cardiac structure and/or function, showing elevated natriuretic peptide levels (BNP>35 ng/L or/and N-terminal pro-BNP >125 ng/L).
3. Have reviewing echocardiography after discharge.

Exclusion Criteria:

1. Patients with hypertrophic, restrictive, or invasive cardiomyopathy and congenital or rheumatic heart disease.
2. Patients with heart transplantation during follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants in the study are HF patients hospitalized in the Department of Cardiology of the First Affiliated Hospital of Harbin Medical University who had no less than two echocardiograms at baseline and during the follow-up period, between January 2014 to December 2022.
Sampling Method: Probability Sample
Enrollment: 422 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-05-20 (Actual)

PRIMARY OUTCOMES:
change of left ventricular ejection fraction | 3 months
  left ventricular ejection fraction value in millimeters

SECONDARY OUTCOMES:
change of clinical predictor of EF improvement | 3 months
  weight in kilograms, height in meters(weight and height will be combined to report BMI in kg/m^2)
the independent clinical predictor of HFimpEF | 3 months
  prealbumin in mg/L

CONTACTS AND LOCATIONS:
Locations (1):
- Yihui Kong, Harbin, Heilongjiang, China